CLINICAL TRIAL: NCT05227638
Title: Investigation of the Efficacy of PNF and Schroth Treatment in Adolescent Idiopathic Scoliosis
Brief Title: Investigation of the Efficacy of PNF and Schroth Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Hanifi Kaya (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Sponsor-Investigator, Mehmet Hanifi Kaya, Lecturer, Kirsehir Ahi Evran Universitesi
Organization: Kirsehir Ahi Evran Universitesi (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: E-10879717-050.01.04-2542
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth group (Active Comparator): The Schroth group performed Schroth exercises
  Interventions: Other: exercise
- PNF group (Active Comparator): PNF group (PG) performed "chop and lift" exercises
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — participants were between ages 10-18, volunteered for the study, were diagnosed with adolescent idiopathic scoliosis, were Cobb angle between 10-30 degrees, were 0-3 Risser sign, and were Lenke curve type 1.
  Other Names: PNF group

SUMMARY:
our study was to compare the advantages of Schroth and PNF methods used in AIS treatment

DETAILED DESCRIPTION:
there are studies showing that Schroth and PNF are effective on AIS seperately. While there are studies showing that Schroth is particularly effective on AIS, the number of studies on PNF is insufficient. However, no evidence was found comparing the efficacy of Schroth and PNF. Therefore, the aim of our study was to compare the advantages of Schroth and PNF methods used in AIS treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants were between ages 10-18
* Volunteered for the study.
* Diagnosed with adolescent idiopathic scoliosis
* Cobb angle between 10-30 degrees
* 0-3 Risser sign
* Lenke curve type 1

Exclusion Criteria:

* non-idiopathic scoliosis
* previous spinal surgery
* who had exercise contraindications who had rheumatological disease who had mental handicap and who another neuromuscular problem

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Cobb angle | 8 week
  anteroposterior x-ray was taken with the entire spine of the patients standing

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Hanifi KAYA, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaya MH, Buyukturan O, Buyukturan B, Alkan H, Erbahceci F. Comparison of the efficacy of the Schroth method and proprioceptive neuromuscular facilitation technique in adolescent idiopathic Scoliosis: a randomized controlled, single-blinded study. J Bodyw Mov Ther. 2025 Sep;43:35-41. doi: 10.1016/j.jbmt.2025.04.003. Epub 2025 Apr 17. PMID 40483147